CLINICAL TRIAL: NCT06012383
Title: A Phase IV, Post Marketing, Prospective, Observational Cohort Study to Investigate Safety and Effectiveness of Alvocade® in Iranian Patients With Multiple Myeloma
Brief Title: Alvocade® (Bortezomib) Safety and Effectiveness Study
Status: Completed | Type: Observational
Sponsor: NanoAlvand (Industry)
Responsible Party: Sponsor
Other Study IDs: BOR.NA.MR.95.IV
Record Dates: First submitted 2023-08-13; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Multiple Myeloma, Refractory
Keywords: Multiple Myeloma; Bortezomib; Safety; Alvocade
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NanoAlvand Bortezomib: 1.3 mg/m2 Bortezomib, IV infusion
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — Alvocade® was given with a dose of 1.3 mg/m2.
  Other Names: Alvocade®

SUMMARY:
This study is a phase IV, post-marketing, observational, cohort study for safety and effectiveness evaluation of Alvocade® use in Iranian patients with multiple myeloma. No control groups were considered in the study design. The primary objective of this study was safety assessment, including the incidence of adverse events (AEs).

DETAILED DESCRIPTION:
This study is a phase IV, post-marketing, observational, cohort study for safety and effectiveness evaluation of Alvocade® use in Iranian patients with multiple myeloma. Data were gathered in two booklets, containing information on sixteen injections, which were filled by the designated physician.

Exposure to Alvocade® in this study was defined as administration of bortezomib (Alvocade®, NanoAlvand) with a dose of 1.3 mg/m2, once every 3 weeks during 2.5 to 5.5 months (16 injections).

The primary objective of this study was safety assessment, including the incidence of adverse events (AEs).

This study was single arm and the sample size of this study was 59 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple myeloma were included in the study.

Exclusion Criteria:

* There were no exclusion criteria for this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A population of 57 Iranian patients diagnosed with multiple myeloma under chemotherapy regimens with Alvocade® (with a dose of 1.3 mg/m2), were enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Safety Assessment | up to 6 months
  Safety assessment, including the incidence of AEs. All AEs were classified based on the Medical Dictionary for Regulatory Activities (MedDRA Desktop Browser 4.0 Beta) terms as System Organ Class (SOC) and Preferred Term (PT). All the reported events were graded according to the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0). Moreover, seriousness of AEs was assessed according to International Council for Harmonisation (ICH-E2B) guidelines. The causality relation was assessed based on the World Health Organization (WHO) criteria.

SECONDARY OUTCOMES:
Effectiveness Assessment | up to 6 months
  Response categories (Stable Disease (SD), Partial Response (PR), Very Good Partial Response (VGPR), Complete Response (CR), and stringent Complete Response (sCR)) were defined and reported based on the uniform response criteria of the International Myeloma Working Group.

CONTACTS AND LOCATIONS:
Overall Officials: Mani Ramzi, Prof., Principal Investigator — Shiraz University of Medical Sciences, Shiraz, Iran